CLINICAL TRIAL: NCT03593135
Title: Effect of Apple Cider Vinegar in Type 2 Diabetic Patients With Poor Glycemic Control: a Randomized Controlled Design
Brief Title: Effect of Apple Cider Vinegar in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Responsible Party: Principal Investigator, Sofia Kausar, Clinical Nutritionist, Sheikh Zayed Federal Postgraduate Medical Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1481
Record Dates: First submitted 2018-06-24; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Randomized Controlled Trial; Diabetes Mellitus
Keywords: vinegar; diabetes; hyperglycemia; hypercholesterolemia; nutraceutical
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Hypercholesterolemia | interventions — Metformin; Methods; Water

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Single-blinded trial, Intervention and placebo given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Intervention group taking their diet according to their original meal pattern only dietary guideline were given regarding high glycaemic and low glycaemic diet. Medical treatments continued (including tablet Tagipment 50mg/1000mg twice a day)(Metformin + Sitagliptin group). 15ml apple cider vinegar (American garden organic vinegar) (containing 5% acetic acid) mixed in 200ml water during meal at night time was prescribed.
  Interventions: Dietary Supplement: Apple Cider Vinegar and tablet Tagipmet (Metformin + Sitagliptin group)
- Comparison group (Placebo Comparator): Control group also taking their diet according to their original meal pattern only dietary guideline were given regarding high glycaemic and low glycaemic diet. Medical treatment continued (including tablet Tagipmet 50mg/1000mg twice a day)( Metformin + Sitagliptin group). Flavor of apple cider vinegar used as placebo, mixed in 200ml plain water during meal at night time.
  Interventions: Other: Water with Apple Cider vinegar flavor and tablet Tagipmet (Metformin + Sitagliptin group)

INTERVENTIONS:
Dietary Supplement: Apple Cider Vinegar and tablet Tagipmet (Metformin + Sitagliptin group) — 15ml apple cider vinegar (American garden organic vinegar) (containing 5% acetic acid) mixed in 200ml water during meal at night time, for 3 months and tablet Tagipmet 50mg/1000mg (Metformin + Sitagliptin group) twice a day. NOTE medical treatment is our inclusion criteria.
  Other Names: intervention
  Arms: Intervention group
Other: Water with Apple Cider vinegar flavor and tablet Tagipmet (Metformin + Sitagliptin group) — Flavor of apple cider vinegar in 200 ml water is added and given to have a placebo effect and tablet Tagipmet 50mg/1000mg (Metformin + Sitagliptin group) twice a day. NOTE medical treatment is our inclusion criteria.
  Other Names: Placebo
  Arms: Comparison group

SUMMARY:
Background: apple cider vinegar is natural traditional health beneficial nutraceutical used for many aliments. Diabetes mellitus (DM) has been considered a globally major health problem and posing health burden on families and health system. Diabetes is associated with life style that leading to reduce physical activities and increased in obesity. For development of diabetes the known mechanism are endocrine disorders which cause impaired insulin secretion, hepatic glucose over production and insulin resistance.

Objective: The aim of current randomized controlled trial was to investigate the effect of apple cider vinegar on glycemic control and biochemical parameters in type 2 diabetic patients with poor glycaemic control.

Material & Methods: 110 type 2 diabetic patients according to inclusion criteria were selected and divided into two groups. Interventional group was given 15 ml apple cider vinegar in 200ml water during meal at night time for 3 months. Before and after HbA1C, fasting lipid profile, fasting blood sugar, anthropometrics and dietary changes were assessed and analyzed using IBM SPSS version 20 through paired sample T-test where needed.

.

DETAILED DESCRIPTION:
A study conducted in pre-diabetic healthy individuals showed significant (p=0.05) reduction in HbA1C, in apple cider vinegar group . Many RCTs of human and animals showed hypolipidemic effects of ACV. Anti obesity effect of apple cider vinegar also found in many studies. There is still lot of work going on and this present study is conducted with an objective to measure the effect of apple cider vinegar on HbA1c, fasting blood glucose, fasting lipid profile and body weight.

METHOD:

STUDY DESIGN AND SETTING

This study was a single-blind, randomized-controlled placebo trial. Trial period was three months from August 15, to November 15, 2017. This study was conducted at a 1050 beded tertiary care, teaching hospital of Lahore, Pakistan. This hospital has high diabetics out-patient turnover as being a reputable center in management of diabetes.

PARTICIPANTS:

Adult patients having type 2 diabetes, of both genders with age range from 30-60 years were included. All having BMI between 20-30, non smoker and non alcoholics and all were on standard medical therapy for diabetes (including Metformin + Sitagliptin group). Patients suffering from known chronic renal disease and history of cardiovascular diseases like stroke, ischemic heart disease and known allergy or intolerance to vinegar, reported by the patient or relative and any kind of acute infection were excluded from study.

The sample size of 110 (55 in each group) was estimated by using 95% confidence level,80% power with expected mean change in HbA1c 0.53% and 0.11% for cases treated with apple vinegar and placebo respectively with a SD of 0.77% (by using power + precision 3.0 software). Assuming a 12.6% non-response rate, RCT started with 126 patients, 63 patients in each group. 16 patients were lost to follow up during study period, so finally statistical analysis was done on 110 patients 55 in each group.

DEPENDENT VARIABLES: A structured questionnaire was used for collecting respondents' information. Blood samples were taken for biochemical test (HbA1c, lipid profile and fasting blood glucose) and anthropometrics measurements were done.

Anthropometric measurements: Height was measured in centimeter to nearest 0.1 cm by using standard stadiometer before intervention and weight was measured in kilogram to nearest 100 g with wearing light cloth by using a calibrated weighing scale machine before and after intervention. Hip/waist ratio and mid upper arm were measured with measuring tape in centimeter to nearest 0.1cm. The BMI of study participants were classified as underweight, normal, over weight and obese according to WHO criteria weight was measured as weight (kg)/height (cm)2.

Biochemical assessments:

At before start of intervention and after intervention 5ml venous blood sample was taken with 12hours fasting for biochemical assessments including blood sugar fasting, HbA1C (glycated hemoglobin), total cholesterol, low density lipoprotein, high density lipoprotein and triglyceride were evaluated.

CONFOUNDING VARIABLES:

Dietary intake:

Diet of study participants can influence and confound the intervention during study period so it was assessed through food frequency questionnaire. Food frequency was filled two times before and after intervention to measure change during study period which can actually confound the effect of apple cider vinegar. The food frequency questionnaire was structured according to Pakistan's cultural food preferences and choices. FFQs contained methods of food preparation, frequency per day and per week and portion size/ amount of food consumed in categories from never, monthly to 1-7 days in a week. Food exchange lists were used to assess the portion size of food. FFQ composed of cereal group, fruits, vegetable, meat, milk, fat/oil, snacks and beverages.

INDEPENDENT VARIABLE/ INTERVENTION: This selected nutraceutical (Apple cider vinegar) was given for three months. Apple cider vinegar was provided to patients and instructions were given to all participants about the uses of apple cider vinegar and strictly follow the prescribed nutraceutical given as per following schedule; Group I: Intervention group Intervention group taking their diet according to their original meal pattern only dietary guideline were given regarding high glycaemic and low glycaemic diet. Medical treatments continued (including Metformin + Sitagliptin group). 15ml apple cider vinegar (American garden organic vinegar) (containing 5% acetic acid) mixed in 200ml water during meal at night time was prescribed.

Group II: comparison group Control group also taking their diet according to their original meal pattern only dietary guideline were given regarding high glycaemic and low glycaemic diet. Medical treatment continued (including Metformin + Sitagliptin group). 15ml apple cider vinegar (flavor of ACV in plan water was used as placebo) mixed in 200ml plain water during meal at night time.

Statistical analysis:

Descriptive statistical analysis was done for demographic profile, categorical and numerical variables by measuring frequency, percentage, mean and standard deviation of all samples. Paired sample T test was used for anthropometrics measurement and biochemical assessment for two time assessment before and after intervention. Independent sample t-test was used for comparison between groups. Where needed ANOVA was also applied. McNemar statistical test was used to assess the food frequency questionnaire before and after intervention.

Ethical considerations:

Proper ethical clearance was obtained from Institutional Review Board of Shaikh Zayed Medical Complex before starting the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients having uncontrolled type 2 diabetes with raised HbA1c levels.
* Both gender.
* Age ranging from 30-60 years.
* All having body mass index between 20-30.
* Non alcoholics.
* Non smoker.
* All were on standard medical therapy for diabetes (including Metformin + Sitagliptin group).

Exclusion Criteria:

* Patients suffering from known chronic renal disease.
* History of cardiovascular diseases like stroke, ischemic heart disease.
* Known allergy to vinegar.
* intolerance to vinegar, reported by the patient or relative.
* Any kind of acute infection were excluded from study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
HbA1c (Glycosylated Hemoglobin) | 3 months
  Before start of intervention and after intervention 5ml venous blood sample was taken for biochemical analysis of HbA1C (glycosylated hemoglobin) in sterilized tubes,commercial kits of Siemens for Dimmension RxL used and the HbA1C measuement is based on a turbidimetric inhibition immunoassay (TINIA) priniciple.

SECONDARY OUTCOMES:
blood sugar fasting | 3 months
  Before start of intervention and after intervention 5ml venous blood sample was taken with 12 hours fasting for biochemical analysis of blood sugar fasting in sterilized dray tubes,commercial kits of Siemens for Dimmension XL and photometric methods for analysis was used.
fasting lipid profile | 3 months
  Before start of intervention and after intervention 5ml venous blood sample was taken with 12 hours fasting for biochemical analysis of fasting lipid profile commercial kits of Rodex for Dimmension Rxl and photometric methods for analysis were used.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaikh Zayed Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke P. Seat belts. Lancet. 1977 May 28;1(8022):1155. doi: 10.1016/s0140-6736(77)92414-x. No abstract available. PMID 68254